CLINICAL TRIAL: NCT06535659
Title: VitaFlow Liberty™ Transcatheter Aortic Valve System Post-market Clinical Follow-up Study
Brief Title: VitaFlow LIBERTY Europe
Status: Recruiting | Type: Observational
Sponsor: Shanghai MicroPort CardioFlow Medtech Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: VitaFlow EU-2024
Record Dates: First submitted 2024-07-21; First posted 2024-08-02 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Aortic Valve Stenosis
Keywords: Transcatheter aortic valve replacement
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single arm clinical investigation
  Interventions: Device: VitaFlow Liberty™ Transcatheter Aortic Valve System

INTERVENTIONS:
Device: VitaFlow Liberty™ Transcatheter Aortic Valve System — Transcatheter Aortic Valve Replacement with VitaFlow Liberty™ Transcatheter Aortic Valve System.
  Patients will receive transcatheter aortic valve replacement and examinations at the screening, procedure, discharge, and follow-up per local standard of care.

SUMMARY:
This is a prospective, single-arm, multi-center, observational, post-market registry to document the clinical safety and performance of MicroPort CardioFlow VitaFlow Liberty™ Transcatheter Aortic Valve System in the routine practice for the treatment of severe aortic valve stenosis. The primary endpoint is the composite rate of all-cause mortality and stroke with disability at 12 months.

Patients will receive transcatheter aortic valve replacement and examinations at the screening, procedure, discharge, and follow-up per local standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of age≥ 18 years
2. Subjects with severe, symptomatic, calcific aortic stenosis who are considered at high risk for surgical aortic valve replacement (AVR).
3. Subject can understand the purpose of the clinical investigation, has signed voluntarily the informed consent form and is agreeing to the scheduled follow up requirements.

Exclusion Criteria:

1. Pre-existing mechanical heart valve in aortic position
2. A known hypersensitivity or contraindication to all anticoagulation /antiplatelet regimens (or inability to be anticoagulated for the index procedure), to nickel or titanium, to nitinol, to dairy products, to polyethylene terephthalate (PET) or contrast media
3. Ongoing sepsis, including active endocarditis
4. Anatomically not suitable for the VitaFlow Liberty TAV system
5. LVEF<20%
6. Estimated life expectancy of less than 12 months
7. Any medical, social or psychological condition that in the opinion of the Heart Team precludes the subject from receiving transcatheter aortic valve replacement
8. Currently participating in another drug or device trial (excluding registries) for which the primary endpoint has not been assessed
9. Inability to comply with the clinical investigation follow-up or other clinical investigation requirements
10. Patients temporally unable to provide written informed consent (e. g. unconscious emergency patients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic, severe calcified aortic stenosis who are at high surgical risk.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2027-06-06 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
Composite rate of all-cause mortality and stroke with disability | 12 months post procedure
  Composite rate of all-cause mortality and stroke with disability

SECONDARY OUTCOMES:
Safety outcomes defined by VARC3 | 30 days, 12 months, and 2-5 years post procedure
  Rate of all-cause mortality, myocardial infarction, stroke, implanted related new and/or worsen conduction disturbances and arrhythmias, new permanent pacemaker implantation, procedure-related or valve-related hospitalization defined by VARC 3.
Safety outcomes defined by VARC3 | 30 days and 12 months post procedure
  Rate of type 2-4 bleeding, major vascular and access-related complications, acute kidney injury (stage 2-4) defined by VARC 3
Safety outcomes defined by VARC3 | acute procedure (within 24 hours)
  Rate of other acute procedural and technical valve related complications: conversion to surgery; unplanned use of mechanical circulatory support; implantation of multiple (>1) transcatheter valves during the index hospitalization; valve mal-position
Device success | 30 days post implantation
  Device success defined by VARC 3
Device early safety | 30 days post implantation
  Device early safety defined by VARC 3
Bioprosthesis haemodynamic function | Discharge (24 hours to 7 days), 30 days,12 months and 2-5 years post implantation
  Bioprosthesis haemodynamic function (assessed by echocardiography) including effective orifice area (cm2).
Bioprosthesis haemodynamic function | Discharge (24 hours to 7 days), 30 days,12 months and 2-5 years post implantation
  Bioprosthesis haemodynamic function (assessed by echocardiography) including mean transvalvular gradient (mmHg).
Bioprosthesis haemodynamic function | Discharge (24 hours to 7 days), 30 days,12 months and 2-5 years post implantation
  Bioprosthesis haemodynamic function (assessed by echocardiography) including aortic regurgitation (paravalvular, central and total).
Bioprosthetic valve dysfunction | 12 months and 2-5 years post procedure
  Moderate or severe haemodynamic valve deterioration defined by VARC3
Bioprosthetic valve dysfunction | 12 months and 2-5 years post procedure
  Bioprosthetic valve failure defined by VARC3
Bioprosthetic valve dysfunction | 12 months and 2-5 years post procedure
  Clinically significant valve thrombosis defined by VARC3
NYHA Classification | From baseline to discharge (24 hours to 7 days), 30 days, 12 months and 2-5 years post procedure
  Changes in cardiac function at discharge, 30 days and 12 months and 2-5 years post implantation according to the NYHA Classification Scheme compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Darren Mylotte, MD, Principal Investigator — Galway University Hospital
Locations (6):
- Galway University Hospital, Galway, Ireland
- Ospedale Cisanello, Pisa, Italy
- Spain (3):
  - Hospital Universitario de a Coruna, A Coruña
  - Hospital Clínico San Carlos, Madrid
  - Hospital clinico Universitario de Valladolid, Valladolid
- Luzerner Kantonsspital | Herzzentrum, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No